CLINICAL TRIAL: NCT03121599
Title: A Study of 18F-FLT Positron Emission Tomography (PET)/Computed Tomography Imaging in Pediatrics With Myeloproliferative Neoplasms
Brief Title: 18F-FLT (PET/CT) in Pediatrics With Myeloproliferative Neoplasms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delayed study materials, poor recruitment
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16294/16
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2019-01

CONDITIONS: Essential Thrombocythemia; Primary Myelofibrosis, Fibrotic Stage; Primary Myelofibrosis, Prefibrotic Stage; Polycythemia Vera
MeSH Terms: conditions — Thrombocythemia, Essential; Primary Myelofibrosis; Polycythemia Vera | interventions — Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 18F-FLT PET/CT (Experimental): Patients undergo 18F-FLT (3'-18Fluoro-3'-deoxy-Lthymidine) PET/CT (Positron Emission Tomography/ Computed Tomography) at baseline. No specific dietary restrictions or hydration are required for FLT-PET scans, however, patients will be urged to drink plenty of water before and after the PET studies. [18F] FLT will be prepared by the cyclotron core facility and assessed for quality control following "good manufacturing practice" criteria. The radiopharmaceutical will immediately be brought to the Molecular Imaging and Therapy Service Radiopharmacy for dispensation in the PET suite. For each scan, patients will receive approximately up to 370 MBq (target of 10 mCi) [18F] FLT by intravenous infusion.
  Interventions: Device: Diagnostic (18F-FLT PET/CT)

INTERVENTIONS:
Device: Diagnostic (18F-FLT PET/CT) — The tracer compound [F-18] FLT will be injected into the patient's veins in a small volume of normal saline solution. The PET scan data collection is started immediately and is continued for 2 hours.
  Other Names: 18F-FLT PET/CT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; Fluorothymidine F 18

SUMMARY:
The Main purpose of this project to study the uptake pattern of FLT-PET and it is value in assessing the malignant hematopoiesis in MPN within the pediatric age group, in terms of diagnosis, staging and monitoring response to therapy. As well as, evaluating FLT-PET as a novel non-invasive technique in cases with MPN and its role in comparison to the standard bone marrow biopsy with regard to disease diagnosis, assessment of disease activity, detection of transformation, monitoring of treatment response and grading of fibrosis.Furthermore, we aim to study the association of FLT-PET uptake patterns with different genetic makeup (JAK2, CALR positive, MPL, or Triple negative disease) or allele burden in cases of Pre-PMF with the ability of FLT-PET to differentiate between Pre-PMF and ET.

Although MPNs are diseases of elderly, MPN is diagnosed in younger age groups in a considerable number of cases. Since most of the available data as well as current WHO classification criteria emphases on the "average" MPN patients who range in age between 55 and 65 years. Less consistent data are available in the groups of patients presenting below this median age, such as children and younger adults which we're planning to reveal.

ELIGIBILITY:
Inclusion Criteria:

* Cases fulfilling WHO (World Health Organization) 2016 diagnostic criteria for MPN including: Chronic myeloid leukemia, BCR-ABL1-positive (BCR-ABL = fusion gene from BCR (breakpoint cluster region gene/BCR gene product), Chronic neutrophilic leukemia (CNL), Polycythemia vera, Primary myelofibrosis prefibrotic/early stage, Primary myelofibrosis overt fibrotic stage, Essential thrombocythemia, Chronic eosinophilic leukemia, not otherwise specified (NOS) and Myeloproliferative neoplasm, unclassifiable.
* Age between 14 and 18 years old
* Patient accepts to sign inform consent
* ECOG (Eastern Cooperative Oncology Group) performance less than or equal 2

Exclusion Criteria:

* Patient not fulfilling the inclusion criteria.
* Vulnerable groups: pregnant, minors, prisoners will not be included.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2017-06-11 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Evaluate the uptake of 3'-deoxy-3'-[18F] fluorothymidine (FLT) positron emission tomography/computed tomography (PET) in children with MPNs | 12 Months
  Evaluate the uptake of 3'-deoxy-3'-[18F] fluorothymidine (FLT) positron emission tomography/computed tomography (PET) imaging and it is value in assessing the malignant hematopoiesis in children with MPNs.

SECONDARY OUTCOMES:
Number of patients who have similar diagnosis and pattern between FLT and Bone Marrow | 12 months
  Assessing of WHO diagnostic criteria for diagnosing MPNs. Measurements would include: Bone marrow cellularity, trilineal assessment, megakaryocytic morphologic characteristics (atypia, clustering, size, lobulation), staging of primary myelofibrosis into prefibrotic/early stage, Primary myelofibrosis and overt fibrotic stage prefibrotic, grade of fibrosis, blast percentage, presence of transformation, intrasinusoidal hematopoiesis, dysplasia (if present).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Yassin, Principal Investigator — Hamad Medical Corporation
Locations (1):
- National Center for Cancer Care & Research (NCCCR), Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pikman Y, Lee BH, Mercher T, McDowell E, Ebert BL, Gozo M, Cuker A, Wernig G, Moore S, Galinsky I, DeAngelo DJ, Clark JJ, Lee SJ, Golub TR, Wadleigh M, Gilliland DG, Levine RL. MPLW515L is a novel somatic activating mutation in myelofibrosis with myeloid metaplasia. PLoS Med. 2006 Jul;3(7):e270. doi: 10.1371/journal.pmed.0030270. PMID 16834459
- [Background] Beer PA, Campbell PJ, Scott LM, Bench AJ, Erber WN, Bareford D, Wilkins BS, Reilly JT, Hasselbalch HC, Bowman R, Wheatley K, Buck G, Harrison CN, Green AR. MPL mutations in myeloproliferative disorders: analysis of the PT-1 cohort. Blood. 2008 Jul 1;112(1):141-9. doi: 10.1182/blood-2008-01-131664. Epub 2008 May 1. PMID 18451306
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Agool A, Schot BW, Jager PL, Vellenga E. 18F-FLT PET in hematologic disorders: a novel technique to analyze the bone marrow compartment. J Nucl Med. 2006 Oct;47(10):1592-8. PMID 17015893
- [Background] Chalkidou A, Landau DB, Odell EW, Cornelius VR, O'Doherty MJ, Marsden PK. Correlation between Ki-67 immunohistochemistry and 18F-fluorothymidine uptake in patients with cancer: A systematic review and meta-analysis. Eur J Cancer. 2012 Dec;48(18):3499-513. doi: 10.1016/j.ejca.2012.05.001. Epub 2012 May 31. PMID 22658807
- [Background] Chen W, Cloughesy T, Kamdar N, Satyamurthy N, Bergsneider M, Liau L, Mischel P, Czernin J, Phelps ME, Silverman DH. Imaging proliferation in brain tumors with 18F-FLT PET: comparison with 18F-FDG. J Nucl Med. 2005 Jun;46(6):945-52. PMID 15937304
- [Background] Ott K, Herrmann K, Schuster T, Langer R, Becker K, Wieder HA, Wester HJ, Siewert JR, zum Buschenfelde CM, Buck AK, Wilhelm D, Ebert MP, Peschel C, Schwaiger M, Lordick F, Krause BJ. Molecular imaging of proliferation and glucose utilization: utility for monitoring response and prognosis after neoadjuvant therapy in locally advanced gastric cancer. Ann Surg Oncol. 2011 Nov;18(12):3316-23. doi: 10.1245/s10434-011-1743-y. Epub 2011 May 3. PMID 21537865
- [Background] Ott K, Rachakonda PS, Panzram B, Keller G, Lordick F, Becker K, Langer R, Buechler M, Hemminki K, Kumar R. DNA repair gene and MTHFR gene polymorphisms as prognostic markers in locally advanced adenocarcinoma of the esophagus or stomach treated with cisplatin and 5-fluorouracil-based neoadjuvant chemotherapy. Ann Surg Oncol. 2011 Sep;18(9):2688-98. doi: 10.1245/s10434-011-1601-y. Epub 2011 Feb 24. PMID 21347786
- [Background] Graf N, Herrmann K, den Hollander J, Fend F, Schuster T, Wester HJ, Senekowitsch-Schmidtke R, zum Buschenfelde CM, Peschel C, Schwaiger M, Dechow T, Buck AK. Imaging proliferation to monitor early response of lymphoma to cytotoxic treatment. Mol Imaging Biol. 2008 Nov-Dec;10(6):349-55. doi: 10.1007/s11307-008-0162-3. Epub 2008 Aug 14. PMID 18704591
- [Background] Leonard JP, LaCasce AS, Smith MR, Noy A, Chirieac LR, Rodig SJ, Yu JQ, Vallabhajosula S, Schoder H, English P, Neuberg DS, Martin P, Millenson MM, Ely SA, Courtney R, Shaik N, Wilner KD, Randolph S, Van den Abbeele AD, Chen-Kiang SY, Yap JT, Shapiro GI. Selective CDK4/6 inhibition with tumor responses by PD0332991 in patients with mantle cell lymphoma. Blood. 2012 May 17;119(20):4597-607. doi: 10.1182/blood-2011-10-388298. Epub 2012 Mar 1. PMID 22383795
- [Background] Zhang CC, Yan Z, Li W, Kuszpit K, Painter CL, Zhang Q, Lappin PB, Nichols T, Lira ME, Affolter T, Fahey NR, Cullinane C, Spilker M, Zasadny K, O'Brien P, Buckman D, Wong A, Christensen JG. [(18)F]FLT-PET imaging does not always "light up" proliferating tumor cells. Clin Cancer Res. 2012 Mar 1;18(5):1303-12. doi: 10.1158/1078-0432.CCR-11-1433. Epub 2011 Dec 14. PMID 22170262
- [Background] Shields AF, Grierson JR, Dohmen BM, Machulla HJ, Stayanoff JC, Lawhorn-Crews JM, Obradovich JE, Muzik O, Mangner TJ. Imaging proliferation in vivo with [F-18]FLT and positron emission tomography. Nat Med. 1998 Nov;4(11):1334-6. doi: 10.1038/3337. PMID 9809561
- [Background] Vesselle H, Salskov A, Turcotte E, Wiens L, Schmidt R, Jordan CD, Vallieres E, Wood DE. Relationship between non-small cell lung cancer FDG uptake at PET, tumor histology, and Ki-67 proliferation index. J Thorac Oncol. 2008 Sep;3(9):971-8. doi: 10.1097/JTO.0b013e31818307a7. PMID 18758298